CLINICAL TRIAL: NCT05773625
Title: Measuring, Analyzing and Mapping Environmental Influences on (and Changes in) Spatial Patterns: Evidence for Just-in-time Adaptive Interventions
Brief Title: JITAIs: Optimization of Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Dr. Laura H.H. Winkens, Researcher and lecturer, Wageningen University and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 555003027
Record Dates: First submitted 2023-01-12; First posted 2023-03-17 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Eating Behavior; Chronic Disease
MeSH Terms: conditions — Feeding Behavior; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group of app (Other): All participants will first use the app one week without receiving just-in-time notifications. Their movement patterns are collected through GPS. In the second week, they will receive just-in-time notifications based on their chosen goal. Participants will act as their own control group.
  Interventions: Device: Just-In-Time Adaptive Intervention

INTERVENTIONS:
Device: Just-In-Time Adaptive Intervention — Participants will be exposed to a new innovative app to test.

SUMMARY:
The goal of this feasibility study is to get insight into the receptivity of a JITAI aimed at healthy dietary intake in inhabitants of a small city in the Netherlands.

The main question it aims to answer is:

• what is the right time and the right location to send notifications to people and for what type of interventions are people most receptive? Furthermore, the aim is to get insight into the relevance and usability of the app, the privacy concerns that people have and the perceived effectiveness of the app on dietary intake.

Participants will test our app for 2 weeks, of which they will receive prompts during one week.

DETAILED DESCRIPTION:
JITAIs have already been developed in the fields of physical activity, smoking, alcohol use and mental illness. Within these fields, results were promising since JITAIs have proven to be effective in changing behaviour. Until now, no JITAIs have been developed that primarily focus on eating behaviour and it is expected that this type of interventions yields great potential in changing eating behaviour.

In this feasibility study a newly developed app is tested with the aim to get insight into what factors influence the receptiveness of people. Receptiveness is the person's ability to receive, process, and use the support provided, which is a prerequisite to achieve behaviour change. In the pilot study the aim is to investigate when and where the right time is to send notifications to people and for what type of interventions people are most receptive.

Participants are inhabitants of Wageningen who will test our app for 2 weeks. In the first week nothing is expected from the participants, but their movement patterns are collected via GPS; the participants are their own control for the Just-In-Time principle. In the second week the participants receive notifications (i.e., a healthy recipe, a tip for the healthier option at a certain location) based on their selected goal (eating more vegetables, eating less meat, less unhealthy snacking). After receiving the notification, participants are asked to answer several questions. At the end of the day, participants are asked to give us more insight in what they like and dislike to receive, at which locations, at what times, how many times a day, and their reasons behind this.

With this data the app can be further developed (co-creation).

The results of the study will be analysed within persons to visualize patterns. A second goal is to test if the movement patterns of participants can be used to objectively measure if interventions are effective in the future. The movement patterns will be analysed with the use of different algorithms, to see if and how movement patterns can say anything about the behaviour of people (stopping, standing still, alter routes). The movement patterns can be linked to received interventions, locations and receptivity.

Within this pilot study, people are not asked to alter their behaviour. Participants do receive notifications that are focused on making healthier eating choices, but the expectation is that this will not lead to behavioural changes within one week. The goal of the study is to get better insight into the best way to respond to the Just-In-Time principle. Participants will receive zero to several notifications a day for a period of 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Open or motivated to improve their eating behaviour (as this is the target group of the final developed app)

  * Older than 18 years old
  * Living in Wageningen
  * Is able to understand and speak Dutch
  * Having an Android phone

Exclusion Criteria:

* Does not have a specific goal to improve eating behaviour

  * Is under 18 years old
  * Does not live in Wageningen
  * Does not speak and/or understand Dutch
  * Does not have an android phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Receptivity | Receptivity is measured during one week, after every prompt
  The receptiveness is measured with short questions after each prompt on whether the prompt is opportune. Questions on receptiveness are send after every prompt during one week (second week of the study). Dependent on how many locations people visit at which they receive a prompt.

SECONDARY OUTCOMES:
Movement patterns | Location is stored every 5 seconds during two weeks.
  Movement patterns are collected within the city of Wageningen using GPS.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University and Research, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No